CLINICAL TRIAL: NCT00153699
Title: Relationship Between Topiramate Use and Ocular Angle Status: A Prospective Pilot Study
Brief Title: Relationship Between Topiramate Use and Ocular Angle Status
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hong Kong Eye Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2004.310; NCT00518063 (obsolete NCT alias)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Glaucoma, Angle-Closure
Keywords: Side effects; Topiramate
MeSH Terms: conditions — Glaucoma, Angle-Closure | interventions — Topiramate

INTERVENTIONS:
Drug: Topiramate

SUMMARY:
We test the hypothesis whether topiramate narrows the angles which may render Asians more likely to suffer from acute angle closure glaucoma.

DETAILED DESCRIPTION:
Topiramate is approved for the treatment of epilepsy and prophylaxis of migraine attacks. There were case reports of acute angle closure glaucoma (AACG) associated with its use. AACG is particularly common in Asians because of a higher prevalence of narrow angle., we test the hypothesis whether topiramate narrows the angles which may render them more likely to suffer from AACG.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18-75 with an indication for starting topiramate.

Exclusion Criteria:

* Patients with known allergy or intolerance to topiramate.
* Recent exposure to topiramate (<3 months).
* Moderate to severe renal failure.
* Known history of renal calculi or hepatic failure
* Inability to give informed consent.
* Pregnant women or women of child-bearing age who do not practise an acceptable means of contraception.
* Patients known to have angle-closure glaucoma.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2004-09; Study Completion 2007-07 (Estimated)

PRIMARY OUTCOMES:
Change(s) in ophthalmic parameters measured at baseline and after 4 weeks of treatment, including: | 4 weeks
best-corrected visual acuity, refraction, Goldmann applanation tonometry, Gonioscopy, dilated fundus examination, | 4 weeks
and ultrasound biomicroscopy of angle and anterior segment. | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dexter YL Leung, MRCS, Principal Investigator — Hong Kong Eye Hospital; Howan Leung, MRCP, Principal Investigator — Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Hong Kong Eye Hospital, Kowloon
  - Prince of Wales Hospital, Shatin